CLINICAL TRIAL: NCT01773057
Title: Effects of the Computerized Decision Support System 'NHGDoc' on Quality of Care: a Cluster Randomized Controlled Trial
Brief Title: Effects of 'NHGDoc' on Quality of Care
Acronym: NHGDoc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHGDoc 2012
Record Dates: First submitted 2012-11-22; First posted 2013-01-23 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: Computerized Decision Support System; Heart failure; Effects on quality of care; Process of care; Patient outcomes
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active decision support (Experimental): Regular NHGDoc domains plus NHGDoc domain heart failure
  Interventions: Other: NHGDoc domain Heart Failure
- Passive decision support (No Intervention): Regular NHGDoc domains

INTERVENTIONS:
Other: NHGDoc domain Heart Failure — Healthcare providers receive patient specific alerts in terms of diagnosing and treatment of patients with heart failure
  Arms: Active decision support

SUMMARY:
The purpose of this study is to determine whether the computerized decision support system 'NHGDoc' is effective in improving quality of primary care in terms of processes of care (e.g. prescribing behavior of physicians) as well as outcomes of care (e.g. hospital admissions, mortality).

DETAILED DESCRIPTION:
Computerized decision support systems are regarded as useful tools to improve quality of care, but their effects are still uncertain. In the Netherlands 'NHGDoc' a computerized decision support system supported by the Dutch College of General Practitioners (NHG) is currently being implemented among more than 1.000 general practices in the Netherlands.

The aim of this study is to evaluate the effects of NHGDoc on quality of care. In addition, we want to gain insight into the barriers and facilitators that affect the systems' impact.

A cluster randomized controlled trial will be conducted among 120 general practices in the Netherlands. Eligible practices will be randomized to receive either the regular NHGDoc modules (control arm) or the regular modules and an additional module on heart failure (intervention arm). The effect evaluation will focus on processes of care (e.g. prescription behavior) as well as on patient outcomes (e.g. hospital admissions, mortality). Additionally, a process evaluation will be conducted, which includes a focus group study and a survey among participating healthcare providers to evaluate the perceived barriers and facilitators to using 'NHGDoc'.

Results of this study will provide insight in the ability of computerized decision support systems and in particular 'NHGDoc' to improve quality of primary care. Whereas the trial focuses on a specific NHGDoc domain - heart failure - we believe our conclusions are relevant to other primary care areas as well, particularly as this study also explores the factors that contribute to the systems' effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* General practices should use the information system MicroHIS X or Promedico ASP
* NHGDoc should be available in the general practices

Exclusion Criteria:

* General practices that do not meet the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Prescribing of ACE-inhibitors/Angiotensin II | One year
  Percentage of patients with heart failure that is prescribed ACE-inhibitors/Angiotensin II
Prescribing of beta blockers | One year
  Percentage of heart failure patients that is prescribed beta blockers
Prescribing of diuretics | One year
  Percentage of heart failure patients that is prescribed diuretics

SECONDARY OUTCOMES:
Hospital admissions | One year
  Number of hospital admissions of patients with heart failure
All cause mortality | One year
  Number of patients with heart failure that die within the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Tijn Kool, PhD, Principal Investigator — IQ healthcare, Radboud University Nijmegen Medical Centre, Nijmegen, the Netherlands
Locations (1):
- Radboud University Nijmegen Medical Centre, IQ healthcare, Nijmegen, Netherlands

REFERENCES:
- [Derived] Lugtenberg M, Pasveer D, van der Weijden T, Westert GP, Kool RB. Exposure to and experiences with a computerized decision support intervention in primary care: results from a process evaluation. BMC Fam Pract. 2015 Oct 16;16:141. doi: 10.1186/s12875-015-0364-0. PMID 26474603
- [Derived] Lugtenberg M, Westert GP, Pasveer D, van der Weijden T, Kool RB. Evaluating the uptake and effects of the computerized decision support system NHGDoc on quality of primary care: protocol for a large-scale cluster randomized controlled trial. Implement Sci. 2014 Oct 17;9:145. doi: 10.1186/s13012-014-0145-5. PMID 25322766